CLINICAL TRIAL: NCT05656235
Title: Renal Retention in High Grade Upper Tract Urothelial Cancer: A Phase II Trial of Enfortumab Vedotin and Pembrolizumab in Patients With Upper Tract Urothelial Cancer (UTUC) Who Are Not Candidates for, or Refuse, Nephroureterectomy
Brief Title: Renal Retention in High Grade Upper Tract Urothelial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2249; IRB00327710 (Other: JHM IRB)
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: High Grade Urothelial Carcinoma; Bladder Cancer; Urothelial Carcinoma Bladder
Keywords: Renal Retention in UTUC; High Grade UTUC; refusing nephroureterectomy; Enfortumab vedotin; Padcev; Pembrolizumab; Keytruda
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enfortumab vedotin with Pembrolizumab (Experimental): The study population will include male and female patients over the age of 18 with high grade UTUC (cN0/xM0) and is ineligible for or refuses definitive radical nephroureterectomy (RNU).
  Enfortumab vedotin will be administered on Days 1 and 8 at 1.25mg/kg of every 3-week cycle by intravenous (IV) infusion given over approximately 30 minutes. Pembrolizumab will be administered on Day 1 at 200mg of every 3-week cycle by IV infusion over approximately 30 minutes. Enfortumab vedotin and Pembrolizumab may be administered for up to total of 35 cycles (approximately 2 years).
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab vedotin 1.25mg/kg on Days 1 and 8 every 3 weeks for up to 35 weeks (each cycle = 21 days)
  Other Names: Padcev
Drug: Pembrolizumab — Pembrolizumab 200mg on Day 1 every 3 weeks for up to 35 weeks (each cycle = 21 days)
  Other Names: Keytruda

SUMMARY:
This trial will evaluate the use of combination pembrolizumab and enfortumab vedotin for patients with high grade non-metastatic (cN0/NxMx, no measurable regional lymph nodes, no metastases) upper tract urothelial cancer (UTUC), preferring to forego standard of care radical nephroureterectomy (RNU) surgery. Currently these patients would not be suitable candidates for neoadjuvant trials, as the patients intention is to forego surgery. The patients are also not candidates for metastatic trials, as the patients have no measurable metastasis. The Investigators hypothesize the combination of pembrolizumab and enfortumab vedotin for patients with high grade cN0/NxMx UTUC deferring RNU will lead to event free survival outcomes similar to that achieved by RNU in a historic dataset.

DETAILED DESCRIPTION:
This single arm phase II trial will evaluate the use of enfortumab vedotin and pembrolozumab for high grade upper tract urothelial cancer patients who are unable or unwilling to undergo standard of care nephroureterectomy.

Enfortumab vedotin IV 1.25 mg/kg days 1,8 and pembrolizumab 200 mg IV will be delivered every 21 days in 20 patients with high grade UTUC cT2-T4N0 (non-metastatic) until disease progression outside of the renal/ureter unit and/or intolerance.

Primary objective is event free survival (EFS), defined as the time to systemic relapse or death. The hypothesis is that the combination of pembrolizumab and enfortumab vedotin for patients with high grade non-metastatic UTUC deferring nephroureterectomy will lead to EFS outcomes similar to that achieved by RNU in historical dataset from the Brady Urologic Institute database (based on a subset of 85 patients with high grade UTUC cT2-T4N0 who underwent surgery without perioperative chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of histologically documented, high grade upper tract urothelial cancer, (UTUC can be diagnosed by direct visualization and biopsy, or by 3 dimensional imaging and positive urine cytology) will be enrolled in this study.
2. Patients must refuse definitive radical nephroureterectomy (RNU), or be medically ineligible for surgery. To be medically ineligible, patients must, in the opinion of the clinical team, be at high risk of complications intra or perioperative which would adversely impact morbidity and mortality, including risk of CKD and ESRD.
3. Subjects must not have received prior systemic therapy for locally advanced or metastatic urothelial carcinoma (in other locations such as the bladder or contralateral ureter or renal pelvis) with the following exceptions:

   1. Subjects who received neoadjuvant chemotherapy with recurrence >12 months from completion of therapy are permitted
   2. Subjects that received adjuvant chemotherapy following cystectomy with recurrence >12 months from completion of therapy are permitted
4. Subjects may have radiographic evidence of N1 disease (Metastasis ≤2 cm in greatest dimension, in a single lymph node)
5. Subjects must be age 18 years or older.
6. Archival tumor tissue will be used for eligibility.
7. Subjects must have an ECOG Performance Status score of 0 or 2
8. Subjects must have adequate hematologic and organ function as defined by the baseline laboratory values in Table 3. Transfusion of red blood cells to meet eligibility criteria is allowed.

   Table 3 - Baseline Laboratory Values

   Hematological:

   ANC: ≥1500/μL Platelets: ≥100,000/μL Hemoglobin: ≥9.0 g/dL or ≥5.6 mmol/L

   Hepatic:

   Total Bilirubin: ≤1.5× ULN AST (SGOT) and ALT (SGPT): No adjustment in the starting dose is required when administering PADCEV to patients with mild hepatic impairment (total bilirubin 1 to 1.5 × ULN and AST any, or total bilirubin ≤ULN and AST >ULN).
9. A female subject of childbearing potential is anyone born female who has experienced menarche and who has not undergone surgical sterilization (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or has not completed menopause. Menopause is defined clinically as 12 months of amenorrhea in a person over age 45 in the absence of other biological, physiological, or pharmacological causes. Female subjects of childbearing potential must meet the following conditions:

   * Agree not to try to become pregnant during the study and for at least 6 months after the final dose of study drug.
   * Must have a negative urine or serum pregnancy test (minimum sensitivity of 25 mIU/mL or equivalent units of beta human chorionic gonadotropin [β-hCG]) within 1 day prior to administration of study drug. Female subjects with false positive results and documented verification of negative pregnancy status are eligible for participation.
   * If heterosexually active, must consistently use highly effective methods of birth control, with a failure rate of less than 1% (as described in Appendix L) starting at screening, throughout the study period, and for at least 6 months after the final dose of study drug.
   * Female subjects must agree not to breastfeed or donate ova starting at screening and throughout the study period, and for at least 6 months after the final dose of study drug.
10. A male subject who can father children is anyone born male who has testes and who has not undergone surgical sterilization (e.g., vasectomy followed by a clinical test proving that the procedure was effective). Male subjects who can father children, must meet the following conditions:

    * Must not donate sperm starting at screening and throughout the study period, and for at least 6 months after the final dose of study drug. Male subjects will be informed about the negative risk to reproductive function and fertility from the study treatment. Prior to treatment male subjects should be advised to seek information on fertility preservation and sperm cryoconservation.
    * Must consistently use highly effective methods of birth control, with a failure rate of less than 1% (as described in Appendix L) starting at screening and continue throughout study period and for at least 6 months after the final dose of study drug.
    * Male subjects with a pregnant or breastfeeding partner(s) must consistently use one of 2 contraception options for preventing secondary exposure to seminal fluid (as described in Appendix L) for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for at least 6 months after the final dose of study drug.
11. Subjects must provide written informed consent.

Exclusion Criteria:

1. Subjects who have previously received enfortumab vedotin or other MMAE-based ADCs.
2. Subjects who have received prior treatment with a PD-(L)-1 inhibitor for any malignancy, including earlier stage UC, defined as a PD-1 inhibitor or PD-L1inhibitor (including, but not limited to, atezolizumab, pembrolizumab, nivolumab, durvalumab, or avelumab).
3. Subjects who have previously received any prior treatment with an agent directed to another stimulatory or co inhibitory T-cell receptor (including but not limited to CD137 agonists, CTLA-4 inhibitors, or OX-40 agonists).
4. Subjects who have received anti-cancer treatment with chemotherapy, biologics, or investigational agents not otherwise prohibited by exclusion criterion 1-3 that is not completed 4 weeks prior to first dose of study treatment (ongoing hormonal/anti hormonal treatment, e.g., for breast cancer, is allowed, provided that the subject is eligible per exclusion criteria 14).
5. Subjects with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
6. Subjects with an estimated life expectancy <12 weeks
7. Subjects with ongoing sensory or motor neuropathy Grade 2 or higher.
8. Subjects with ongoing clinically significant toxicity associated with prior treatment (including radiotherapy or surgery) that has not resolved to ≤ Grade 1 or returned to baseline.
9. Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of treatment initiation. Routine antimicrobial prophylaxis is permitted.
10. Subjects who have known active hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] detected) infection, testing for hepatitis B and hepatitis C is required if mandated by country health authority. Subjects who have been curatively treated for hepatitis C infection are permitted if they have documented sustained virologic response of 12 weeks.
11. Has a known history of human immunodeficiency virus (HIV) infection. Testing is not required unless mandated by the local health authority.
12. Subjects with conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease. Physiologic replacement doses of corticosteroids are permitted for subjects with adrenal insufficiency.
13. Subjects with another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer. Subjects that have completed all necessary therapy and are considered to be at less than 30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment.
14. Patients may have a history of resected urothelial cancer of the bladder or contralateral upper tract, (including neoadjuvant chemotherapy) in the following categories. These disease states are not exclusions and patients with this history will have this recorded and be considered for study on a case by case basis:

    * pT0, Tis, or T1N0 and have no evidence of disease (NED) for more than 2 years from surgery or chemotherapy;
    * pT2-3aN0 and NED for more than 3 years from surgery or chemotherapy; or
    * >pT3b, or N+ and NED for more than 5 years from surgery or chemotherapy.
    * Patients with concomitant HG UTUC bilaterally will be considered for protocol on a case by case basis.
15. Subjects with a documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with NYHA Class IV within 6 months prior to treatment initiation (Appendix D).
16. Subjects who have received radiotherapy within 2 weeks prior to treatment initiation. Subject must have recovered adequately from the toxicity from the intervention prior to starting study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
17. Subjects who have received major surgery within 4 weeks prior to treatment initiation. Subject must have recovered adequately from complications from the intervention prior to starting study treatment.
18. Subjects with known severe (≥ Grade 3) hypersensitivity to any enfortumab vedotin excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20). Subjects with known severe (≥ Grade 3) hypersensitivity to any pembrolizumab excipient contained in the drug formulations of pembrolizumab. Subjects with known severe (≥ Grade 3) hypersensitivity to the platinum agent selected by the investigator for study treatment. Subjects with known severe (≥ Grade 3) hypersensitivity to the gemcitabine.
19. Subjects with active keratitis or corneal ulcerations. Subjects with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
20. History of autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

    1. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
    2. Brief (<7 days) use of systemic corticosteroids is allowed when use is considered standard of care.
    3. Subjects with vitiligo, psoriasis, type 1 diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy will not be excluded.
    4. Subjects requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded.
    5. Subjects with hypothyroidism that is stable with hormone replacement or Sjögren's syndrome will not be excluded.
21. Subjects with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
22. Subjects who have received a prior allogeneic stem cell or solid organ transplant.

    Subjects who have received a live vaccine or live-attenuated vaccine within 30 days prior to treatment initiation. Administration of killed vaccines is allowed.

    Note: Any licensed COVID-19 vaccine (including for Emergency Use) in a particular country is allowed in the study as long as they are mRNA vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy. Investigational vaccines (i.e., those not licensed or approved for Emergency Use) are not allowed.
23. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
24. Subjects with active tuberculosis
25. Subjects with another underlying medical condition that, in the opinion of the investigator, would impair the ability of the subject to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | 12 months
  Time to relapse or death based on 12 months.

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Baseline, 12 months
  Change from baseline GFR to GFR 1 yr post enrollment

OTHER OUTCOMES:
To evaluate safety and tolerability of the combination of enfortumab vedotin and pembrolizumab | 25 months
  Number of participants experiencing dose limiting toxicities and treatment-related adverse events, as defined by Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Progression free survival | 48 months
  Number of participants without disease recurrence
Overall Survival | 48 months
  Number of participants alive end of trial.
To assess feasibility of obtaining tumor for DNA sequencing including, FGFR mutation / fusion status, from UTUC biopsy specimens | 24 months
  Number participants with tumor available for DNA sequencing including, FGFR mutation / fusion status, from UTUC biopsy specimens
To assess feasibility of obtaining immune biomarker data from UTUC biopsy specimens | 24 months
  Number of participants with immune biomarker data available from UTUC biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Jean Hoffman-Censits, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University: Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No